CLINICAL TRIAL: NCT07046494
Title: A Phase 2, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of RAP-219 for the Acute Treatment of Manic Episodes, With or Without Mixed Features, Associated With Bipolar I Disorder
Brief Title: Study Evaluating the Efficacy and Safety of RAP-219 in Adult Participants With Bipolar I Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rapport Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP-219-BPM-201
Record Dates: First submitted 2025-05-30; First posted 2025-07-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Bipolar 1 Disorder
Keywords: Bipolar; Mania; Acute; In-patient; Manic State; Manic Episode; Mixed Features; Episode with Mixed Features; Mixed Mania; Bipolar Episode
MeSH Terms: conditions — Mania

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled trial of active drug versus placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): Treatment with RAP-219
  Interventions: Drug: RAP-219
- Placebo (Placebo Comparator): Inert comparator matching the active treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RAP-219 — RAP-219 tablets administered orally, once daily for 21 days
  Arms: Active Arm
Other: Placebo — Matching placebo tablets administered orally, once daily for 21 days
  Arms: Placebo

SUMMARY:
This is a clinical research study for an investigational drug called RAP-219 in participants with bipolar I disorder. This study is being conducted to determine if RAP-219 is safe and effective in participants experiencing mania associated with bipolar I disorder.

DETAILED DESCRIPTION:
This is a Phase 2, proof-of-concept, multi-center, randomized, double blind, placebo-controlled study designed to evaluate the efficacy, safety and tolerability of RAP-219 in adult participants experiencing mania associated with bipolar I disorder. This is a 3-week inpatient clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of bipolar I disorder, with or without psychotic symptoms, as confirmed by the Structured Clinical Interview for DSM-5, Clinical Trials Version (SCID-5-CT). Episode may contain mixed features, as confirmed by Montgomery-Åsberg Depression Rating Scale (MADRS).
* Had at least one prior documented manic episode (with or without psychotic symptoms) that required treatment, within 5 years prior to Visit 1

Exclusion Criteria:

* History of any of the following diagnoses: a. schizophrenia; schizoaffective disorder; major depressive disorder; moderate or severe substance or alcohol use disorder; as assessed by the SCID-5-CT b. delirium, dementia, amnestic, or other cognitive disorders; borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorders; by medical history and/or Investigator opinion Note: Any other current diagnoses must be discussed with the Medical Monitor.
* Rapid cycler, defined as experiencing ≥4 distinct mood episodes (ie, manic or depressive) each meeting full DSM-5 criteria in the previous 12 months, and each separated by ≥2 months of full or partial remission, or a switch to an episode of the opposite polarity, as assessed by the SCID-5-CT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS) | Baseline to End of Treatment at Week 3
  The YMRS is a clinician administered scale that consists of 11 items used to assess the severity of manic symptoms (total scores range from 0 to 60). The higher the YMRS score, the more severe the subject's symptoms of mania.

SECONDARY OUTCOMES:
Clinical Global Impression-Bipolar Version (CGI-BP) Severity of Illness Mania score | Baseline to end of Treatment at Week 3
  The CGI-BP Severity of Illness Mania score is a clinician-rated scale used to assess the severity of manic symptoms, depression and overall illness severity in individuals with bipolar disorder. The mania score ranges from 1 (not ill) to 7 (very severely ill), with higher scores indicating greater severity of manic symptoms.
Treatment Emergent Adverse Events (TEAEs) | Baseline to end of Study Period 8 Weeks after date of last dose
  Incidence and severity of treatment-emergent adverse events (TEAEs).
Heart Rate | Baseline to end of Study Period 8 Weeks after date of last dose
  Change in Heart Rate (BPM)
Respiratory Rate | Baseline to end of Study Period 8 Weeks after date of last dose
  Change in Respiratory Rate (breaths per minute)
Body Temperature | Baseline to end of Study Period 8 Weeks after date of last dose
  Change in body temperature
Blood Pressure | Baseline to end of Study Period 8 Weeks after date of last dose
  Change in blood pressure (Hg mm)
Laboratory Analytes | Baseline to end of Study Period 8 Weeks after date of last dose
  Change in laboratory analytes (absolute value)
Electrocardiogram (ECG) QTc interval | Baseline to end of Study Period 8 Weeks after date of last dose
  Changes in electrocardiogram (ECGs); QTc prolongation
Electrocardiogram (ECG) abnormal findings | Baseline to end of Study Period 8 Weeks after date of last dose
  Shift table of normal to abnormal ECG findings
Suicidality | Baseline to end of Study Period 8 Weeks after date of last dose
  Incidence of suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS).

CONTACTS AND LOCATIONS:
Overall Officials: Edwin A Gomez, MD, Principal Investigator — CenExel Research Centers of America
Locations (22):
- United States (22):
  - Pillar Clinical Research - Little Rock, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Inland Psychiatric Medical Group - Chino, Chino, California
  - Synergy Clinical Research Center - San Diego, Lemon Grove, California
  - Collaborative Neuroscience Research - Los Alamitos, Los Alamitos, California
  - NRC Research Institute - Orange, Orange, California
  - CNRI - San Diego, LLC, San Diego, California
  - NeuroBehavioral Hospitals of the Palm Beaches - South, Boynton Beach, Florida
  - United Research Institute, Hialeah, Florida
  - CenExel - Hollywood, Hollywood, Florida
  - Segal Trials - Miami Lakes Medical Research Early Phase, Inpatient & Outpatient Site, Miami Lakes, Florida
  - Neuroscience Research Institute at Ambrosia, West Palm Beach, Florida
  - CenExel - Decatur, Decatur, Georgia
  - Pillar Clinical Research - Chicago, Chicago, Illinois
  - CenExel - Gaithersburg, Gaithersburg, Maryland
  - Arch Clinical Trials, St Louis, Missouri
  - Richmond Behavioral Associates, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Community Clinical Research, Inc., Austin, Texas
  - HD Research - Memorial Hermann Village, Houston, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No